CLINICAL TRIAL: NCT06423235
Title: Efficacy and Safety of Prunella Oral Liquid in the Treatment of Thyroid Nodules: a Multicenter, Prospective, Randomized, Double-blind, Placebo-controlled Study
Brief Title: Efficacy and Safety of Prunella Oral Liquid in the Treatment of Thyroid Nodules
Acronym: ESPTTN
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xintian Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: XK-22-A-002-YJ-002
Record Dates: First submitted 2024-04-07; First posted 2024-05-21 (Actual); Last update posted 2024-05-21 (Actual); Status verified 2024-05

CONDITIONS: Thyroid Nodule
MeSH Terms: conditions — Thyroid Nodule

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- placebo regular dose group (Placebo Comparator)
  Interventions: Drug: regular dose of placebo
- placebo 2x regular dose group (Placebo Comparator)
  Interventions: Drug: 2x regular dose of placebo
- regular dose group of Prunella oral liquid group (Active Comparator)
  Interventions: Drug: regular dose of JiRui® Prunella oral liquid
- 2x regular dose group of Prunella oral liquid group (Active Comparator)
  Interventions: Drug: 2x regular dose of JiRui® Prunella oral liquid

INTERVENTIONS:
Drug: regular dose of JiRui® Prunella oral liquid — Take 10ml twice a day
  Arms: regular dose group of Prunella oral liquid group
Drug: 2x regular dose of JiRui® Prunella oral liquid — Take 20ml twice a day
  Arms: 2x regular dose group of Prunella oral liquid group
Drug: regular dose of placebo — Take 10ml twice a day
  Arms: placebo regular dose group
Drug: 2x regular dose of placebo — Take 20ml twice a day
  Arms: placebo 2x regular dose group

SUMMARY:
A multicenter, prospective, randomized, double-blind, placebo-controlled clinical trial was designed to evaluate the efficacy and safety of Prunella oral liquid in patients with benign thyroid nodules, which belongs to the post-marketing reevaluation clinical study.

In this study, 426 subjects will be enrolled by competitive enrollment at several research centers across China. The main inclusion criteria are:

① Thyroid ultrasound examination found thyroid nodules, can be accompanied by goiter, and the nodules meet the following conditions: 1) There were dominant nodules in single or multiple nodules (the largest diameter of the second largest nodules was not more than 50% of the largest nodules), 2) solid nodules, 3) the longest diameter of nodules was ≥1cm and < 3cm, 4) C-TIRADS 3~4A nodules.

② Patients who met the puncture indication were confirmed by fine needle aspiration biopsy (FNAB) as benign nodules (Bethesda II).

③ Levels of TSH, FT3 and FT4 were normal, and the antibody titers of TgAb and TPOAb were normal.

Eligible subjects will be randomly assigned on a 1:1:2:2 scale to: Group A (placebo conventional dose group, 10 mL/times, 2 times/day), group B (placebo 2x dose group, 10ml/times, 2 times/day), group C (conventional dose group of Prunella oral liquid), group D (Prunella oral liquid 2x dose group). All subjects will receive the treatment for 9 months and follow up at 3rd, 6th, 9th and 12th month.

The primary efficacy endpoint of this study was the rate of change in thyroid nodule volume from baseline at 6 months of treatment. The rate of change in thyroid nodule volume from baseline at 3 and 9 months of treatment was a secondary efficacy endpoint. Other secondary efficacy endpoints included maximum thyroid nodule diameter, number of thyroid nodules, proportion of patients with reduced thyroid nodule volume or ≥50% from baseline, thyroid volume, thyroid function (serum TSH, FT3, FT4, thyroid egg levels (Tg), thyroid antibody levels (TgAb, TPOAb), quality of life evaluation (SF-36), etc. Safety endpoints included incidence of AE/ serious adverse events (SAE), causality, and outcomes. Incidence of AE/SAE leading to discontinuation. Changes in safety laboratory test values from baseline.

ELIGIBILITY:
Inclusion Criteria:

* 18 years old ≤65 years old;
* Thyroid ultrasonography found thyroid nodules, may be accompanied by goiter, and the nodules meet the following conditions: 1) single nodules, or dominant nodules in multiple nodules (the largest diameter of the second largest nodules does not exceed 50% of the largest nodules), 2) solid nodules, 3) the longest diameter of nodules ≥1cm and < 3cm, 4) C-TIRADS 3~4A nodules;
* Patients who met the puncture indications were confirmed by fine needle aspiration biopsy (FNAB) as benign nodules (Bethesda Class II);
* Serum TSH, free thyroid hormone (FT3, FT4) levels were normal, anti-thyroglobulin (TgAb) and anti-thyroid peroxidase (TPOAb) antibody titers were normal;
* Meet the diagnostic criteria of thyroid nodules in TCM;
* Sign the informed consent.

Exclusion Criteria:

* Exclude the patients with Deficiency of Yang syndrome, and the following two conditions can be diagnosed: Shortness of breath, abdominal pain and diarrhea, diarrhea with undigested food, Insufficiency with chills, exhaustion and lethargy, pale tongue and white fur, deep and weak pulse
* Those who have reproductive needs during pregnancy, lactation and within the last 12 months;
* Patients with high possibility of thyroid cancer indicated by ultrasonic signs and malignant confirmed by fine needle biopsy;
* Patients who meet the indications for thyroid nodule surgery, such as local compression symptoms obviously related to the nodule, the tumor is located behind the sternum or in the mediastinum, or strongly require surgery due to appearance or ideological concerns affecting normal life;
* Patients who have taken prunella preparations or other similar Chinese medicines to treat the disease within the past 1 month; Patients using glucocorticoids in the last 3 months;
* Patients who have had or plan to take thyroid hormone, iodine compound, or antithyroid drug therapy during the study period;
* Patients who have previously or plan to undergo ablation, neck radiation, surgery and other non-drug treatments during the study period;
* Patients with parathyroid tumor (PTA), medullary thyroid cancer (MTC) or other malignant tumors, or patients with serious cardiovascular disease, liver and kidney disease, osteoporosis, or patients with a history of mental illness;
* Patients with a family history of thyroid cancer or thyroid cancer syndrome;
* Laboratory test index ALT, AST > 1.5 times the upper limit of reference value or blood creatinine (Scr) > the upper limit of reference value;
* Persons who are known to be allergic to the investigational drug or its ingredients;
* Other patients determined by the investigator to be unsuitable for participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 426 (Estimated)
Dates: Start 2024-07-30 (Estimated); Primary Completion 2025-07-30 (Estimated); Study Completion 2028-07-30 (Estimated)

PRIMARY OUTCOMES:
Rate of change in thyroid nodule volume from baseline at 6 months of treatment. | 180 ± 10 days

SECONDARY OUTCOMES:
Rate of change in thyroid nodule volume from baseline at 3 months of treatment. | 90 ± 7 days.
Rate of change in thyroid nodule volume from baseline at 9 months of treatment. | 270 ± 14 days.
Rate of change in thyroid nodule volume from baseline at 12 months of treatment. | 360 ± 14 days.
The change value of the maximum diameter of thyroid nodules from baseline at 3 months of treatment. | 90 ± 7 days
The change value of the maximum diameter of thyroid nodules from baseline at 6 months of treatment. | 180 ± 10 days
The change value of the maximum diameter of thyroid nodules from baseline at 9 months of treatment. | 270 ± 14 days
The change value of the maximum diameter of thyroid nodules from baseline at 12 months of treatment. | 360 ± 14 days
Proportion of patients with reduced thyroid nodule volume from baseline at 3 months of treatment. | 90 ± 7 days
Proportion of patients with reduced thyroid nodule volume from baseline at 6 months of treatment. | 180 ± 10 days
Proportion of patients with reduced thyroid nodule volume from baseline at 9 months of treatment. | 270 ± 14 days
Proportion of patients with reduced thyroid nodule volume from baseline at 12 months of treatment. | 360 ± 14 days
Proportion of patients with reduced thyroid nodule volume ≥50% from baseline at 3 months of treatment. | 90 ± 7 days
The proportion of patients with reduced thyroid nodule volume ≥50% from baseline at 6 months of treatment. | 180 ± 10 days
Proportion of patients with reduced thyroid nodule volume ≥50% from baseline at 9 months of treatment. | 270 ± 14 days
Proportion of patients with reduced thyroid nodule volume ≥50% from baseline at 12 months of treatment. | 360 ± 14 days
Changes in the number of thyroid nodules from baseline at the 3 months of treatment. | 90 ± 7 days
Changes in the number of thyroid nodules from baseline at the 6 months of treatment. | 180 ± 10 days
Changes in the number of thyroid nodules from baseline at the 9 months of treatment. | 270 ± 14 days
Changes in the number of thyroid nodules from baseline at the 12 months of treatment. | 360 ± 14 days
Proportion of patients with thyroid nodule progression (greater than 50% in volume or greater than 20% in at least 2 diameters from baseline) at 3 months of treatment. | 90 ± 7 days
Proportion of patients with thyroid nodule progression (greater than 50% in volume or greater than 20% in at least 2 diameters from baseline) at 6 months of treatment. | 180 ± 10 days
Proportion of patients with thyroid nodule progression (greater than 50% in volume or greater than 20% in at least 2 diameters from baseline) at 9 months of treatment. | 270 ± 14 days
Proportion of patients with thyroid nodule progression (greater than 50% in volume or greater than 20% in at least 2 diameters from baseline) at 12 months of treatment. | 360 ± 14 days
Rate of change in thyroid volume from baseline at 3 months of treatment. | 90 ± 7 days
Rate of change in thyroid volume from baseline at 6 months of treatment. | 180 ± 10 days
Rate of change in thyroid volume from baseline at 9 months of treatment. | 270 ± 14 days
Rate of change in thyroid volume from baseline at 12 months of treatment. | 360 ± 14 days
Changes in serum TSH, FT3 and FT4 from baseline at the months of treatment. | 90 ± 7 days
Changes in serum TSH, FT3 and FT4 from baseline at the months of treatment. | 180 ± 10 days
Changes in serum TSH, FT3 and FT4 from baseline at 9 months of treatment. | 270 ± 14 days
Changes in serum TSH, FT3 and FT4 from baseline at 12 months of treatment. | 360 ± 14 days
Changes in Tg, TgAb and TPOAb levels from baseline at the 6th month of treatment. | 180 ± 10 days
Proportion of patients with normal thyroid function at 3 months of treatment. | 90 ± 7 days
Proportion of patients with normal thyroid function at 6 months of treatment. | 180 ± 10 days
Proportion of patients with normal thyroid function at 9 months of treatment. | 270 ± 14 days
Proportion of patients with normal thyroid function at 12 months of treatment. | 360 ± 14 days
Subjects' quality of life scores (SF-36) at 3 months of treatment. | 90 ± 7 days
Subjects' quality of life scores (SF-36) at 6 months of treatment. | 180 ± 10 days
Subjects' quality of life scores (SF-36) at 9 months of treatment. | 270 ± 14 days
Subjects' quality of life scores (SF-36) at 12 months of treatment. | 360 ± 14 days

CONTACTS AND LOCATIONS:
Locations (22):
- China (22):
  - Second Hospital of Army Military Medical University, Chongqing, Chongqing Municipality
  - Xiamen Hospital of Traditional Chinese Medicine, Xiamen, Fujian
  - People's Hospital of Guangdong Province, Guangzhou, Guangdong
  - Shenzhen Hospital of Peking University, Shenzhen, Guangdong
  - Shunde Hospital of Southern Medical University, Shunde, Guangdong
  - Wuhan First Hospital, Wuhan, Hubei
  - Jiangsu Province Hospital of Integrated Chinese and Western Medicine, Nanjing, Jiangsu
  - Xuzhou Medical University Hospital, Xuzhou, Jiangsu
  - The Second Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Hospital of Liaoning University of Chinese Medicine, Shenyang, Liaoning
  - People's Hospital of Liaoning Province, Shenyang, Liaoning
  - The First Hospital of Qingdao University, Qingdao, Shandong
  - Weifang People's Hospital, Weifang, Shandong
  - Weihai Hospital, Weihai, Shandong
  - Ruijin Hospital Luwan Branch, Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality
  - Shanghai 10th People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai First People's Hospital, Shanghai, Shanghai Municipality
  - Shanghai Pudong Zhoupu Hospital, Shanghai, Shanghai Municipality
  - First People's Hospital of Yunnan Province, Kunming, Yunnan
  - The First Hospital of Kunming Medical University, Kunming, Yunnan
  - Zhejiang Province Hospital of Integrated Chinese and Western Medicine, Hangzhou, Zhejiang